CLINICAL TRIAL: NCT03699332
Title: A Phase I/II Study to Evaluate the Safety and Feasibility of Multi-modality Imaging Using Indium-111-DOTA-labetuzumab-IRDye800CW in Patients With Peritoneal Carcinomatosis of Colorectal Origin
Brief Title: Multi-modality Imaging in Peritoneal Carcinomatosis of Colorectal Origin
Acronym: MMIPC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL57505.091.16
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Peritoneal Carcinomatosis; Colorectal Cancer; Carcinoma; Neoplasms; Gastrointestinal Cancer
Keywords: image guided surgery; CRS; HIPEC; Fluorescence; Antibodies, monoclonal
MeSH Terms: conditions — Peritoneal Neoplasms; Colorectal Neoplasms; Carcinoma; Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative multi-modality imaging (Experimental): Patients receive a single intravenous dose of Indium-111-DOTA-Labetuzumab-IRDye800CW. At day 4 or 5 after antibody injection a SPECT/CT scan will be acquired. At day 6 or 7 standard of care cytoreductive surgery will be performed. This will be extended with the use of dual-modality imaging.
  Interventions: Drug: Indium-111-DOTA-Labetuzumab-IRDye800CW injection; Radiation: SPECT/CT scan; Procedure: CRS extended with dual-modality imaging

INTERVENTIONS:
Drug: Indium-111-DOTA-Labetuzumab-IRDye800CW injection — Tracer injection
Radiation: SPECT/CT scan — Abdominal and thoracic SPECT/CT scan.
Procedure: CRS extended with dual-modality imaging — cytoreductive surgery will be performed extended with the use of dual-modality imaging.

SUMMARY:
Intraoperative tumor localization and resection can be enhanced using intraoperative fluorescence imaging and radiodetection. Labetuzumab specifically recognizes CEA which is is expressed on > 95% of colorectal cancers.. Therefore Indium-111-DOTA-labetuzumab-IRDye800CW is a perfect dual-labeled antibody for dual-modality image-guided surgery in peritoneal carcinomatosis of colorectal cancer.

DETAILED DESCRIPTION:
In oncologic surgery complete tumor resection is important for treatment outcome and patient survival. When performing cytoreductive surgery (CRS) for peritoneal carcinomatosis of colorectal origin it can sometimes be difficult to distinguish tumor deposits from adhesions and scar tissue. Intraoperative tumor localization and resection can be enhanced using intraoperative imaging techniques (e.g. targeted radioguided or fluorescence guided surgery). A powerful synergy can be achieved by combining radiotracers (e.g. Indium-111) and optical tracers (e.g. IRDye 800CW) conjugated to an antibody against a tumor-associated antigen. Labetuzumab specifically recognises CEA which is expressed on > 95% of all colorectal cancers. Therefore Indium-111-DOTA-labetuzumab-IRDye800CW is a perfect dual-labeled antibody for dual-modality image-guided surgery in peritoneal carcinomatosis of colorectal origin. The concept has been shown in preclinical studies with mice and the investigators will translate this to the clinic.

Eligible patients with peritoneal carcinomatosis of colorectal origin scheduled for CRS + HIPEC will receive dual-labeled labetuzumab 6-7 days before surgery. At day 4 or 5 a SPECT/CT of the abdomen and thorax will be obtained. Cytoreductive surgery at day 7 will be extended with the use of a near-infrared fluorescence camera and a gamma probe.

The aim of this study is to assess the feasibility and safety of intraoperative dual-modality imaging with Indium-111-DOTA-labetuzumab-IRDye800CW in peritoneal carcinomatosis of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of peritoneal carcinomatosis of colorectal origin
* Scheduled for cytoreductive surgery and HIPEC.
* Age over 18 years
* Signed informed consent

Exclusion Criteria:

* Any medical condition present that in the opinion of the investigator will affect patients clinicals status
* Administration of a radionuclide within 10 physical half-lives prior to study enrollment
* Pregnancy or lactation
* Patients with very high (>500ng/ml serum CEA levels
* Known CEA negative tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Fluorescent signal at time of surgery | During cytoreductive surgery
  Can the tumor be identified by the fluorescent signal? Yes/No. Can the tumor be distinguished from normal tissue? Yes/No

SECONDARY OUTCOMES:
Safety of dual-labeled antibody (labetuzumab) as assessed by the number of participants with grade 3 or 4 Adverse Events according to CTCAE v4.0 | 4 weeks
  Safety of dual-labeled antibody injection as assessed by the number of participants with grade 3 or 4 Adverse Events according to CTCAE v4.0
Blood levels of the dual-labeled antibody | 60, 120 and 180 minutes after injection and 4 and 7 days after injection
  Blood samples will be measured for radioactivity in a gamma counter at different timepoints after injection. This will be expressed as percentage injected dose per gram (%ID/g)
Optimal dose of the dual-labeled antibody preparation | 4 weeks
  Optimal dose of dual-labeled antibody for dual modality image guided surgery

CONTACTS AND LOCATIONS:
Overall Officials: JHW de Wilt, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Gooyer JM, Elekonawo FMK, Bremers AJA, Boerman OC, Aarntzen EHJG, de Reuver PR, Nagtegaal ID, Rijpkema M, de Wilt JHW. Multimodal CEA-targeted fluorescence and radioguided cytoreductive surgery for peritoneal metastases of colorectal origin. Nat Commun. 2022 May 12;13(1):2621. doi: 10.1038/s41467-022-29630-9. PMID 35551444